CLINICAL TRIAL: NCT02626338
Title: Pilot Study of Crenolanib Combined With Standard Salvage Chmetherapy in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Pilot Study of Crenolanib Combined With Standard Salvage Chemotherapy in Subjects With R/R AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARO-011
Record Dates: First submitted 2015-11-18; First posted 2015-12-10 (Estimated); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — crenolanib; Mitoxantrone; Cytarabine; Etoposide; etoposide phosphate; fludarabine; fludarabine phosphate; Granulocyte Colony-Stimulating Factor; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): * Mitoxantrone
  * Cytarabine
  * Crenolanib
  Interventions: Drug: Crenolanib; Drug: Mitoxantrone; Drug: Cytarabine
- Arm B (Experimental): * Fludarabine
  * Cytarabine
  * G-CSF
  * Idarubicin
  * Crenolanib
  Interventions: Drug: Crenolanib; Drug: Cytarabine; Drug: Fludarabine; Drug: G-CSF; Drug: Idarubicin
- Arm C (Experimental): * Mitoxantrone
  * Etoposide
  * Cytarabine
  * Crenolanib
  Interventions: Drug: Crenolanib; Drug: Mitoxantrone; Drug: Cytarabine; Drug: Etoposide

INTERVENTIONS:
Drug: Crenolanib
Drug: Mitoxantrone
  Arms: Arm A; Arm C
Drug: Cytarabine
  Other Names: cytosine arabinoside
Drug: Etoposide
  Other Names: Etoposide phosphate
  Arms: Arm C
Drug: Fludarabine
  Other Names: Fludarabine monophosphate
  Arms: Arm B
Drug: G-CSF
  Arms: Arm B
Drug: Idarubicin
  Arms: Arm B

SUMMARY:
The proposed study is designed to combine crenolanib with standard salvage chemotherapy to treat patients with R/R AML irrespective the FLT3 status.

DETAILED DESCRIPTION:
Open label, dose de-escalation, pilot trial of crenolanib with standard salvage chemotherapy. Subjects may receive up to 2 cycles of induction with standard salvage chemotherapy followed by crenolanib. Each arm will enroll approximately 24 patients (72 total); stratification to each arm will be per physician's choice

ELIGIBILITY:
Inclusion Criteria

1. Confirmed diagnosis of AML, including treatment-related secondary AML (except prior MDS) according to World Health Organization (WHO) 2008 classification at treating institution
2. Subjects who are refractory* or who have relapsed** following first line AML therapy with cytarabine/anthracycline based chemotherapy, with or without a tyrosine kinase inhibitor. *Refractory to induction therapy is defined as never achieving CR, CRi or CRp (according to International Working Group criteria) after one line of intensive regimen for AML (re-induction, consolidation and/or transplant allowed) including at least one cytarabine containing induction block with a total dose no less than 700mg/m² per cycle and 3 days of an anthracycline with or without a TKI.

   or

   **First relapse is defined as untreated hematologic relapse (according to International Working Group criteria) after one line of intensive regimen for AML (re-induction, consolidation and/or transplant allowed) including at least one cytarabine containing induction block with a total dose no less than 700mg/m² per cycle and 3 days of an anthracycline with or without a TKI that induced a CR/CRi/CRp. Subjects are allowed to receive induction, consolidation, transplant and/or maintenance prior to achieving their first CR/CRi/CRp.
3. Subjects considered eligible for intensive chemotherapy
4. ECOG performance status ≤ 2
5. Age ≥ 18 years
6. Adequate liver function within 72 hours of enrollment, defined as:

   * Normal total serum bilirubin
   * ALT and AST ≤ 2.0 x ULN
7. Adequate renal function, defined as serum creatinine ≤ 1.5x ULN
8. Women of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 72 hours prior to enrollment "Woman of childbearing potential" is defined as any woman who has not undergone a hysterectomy and who has had menses at any time in the preceding 24 consecutive months
9. Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control (IUD, tubal ligation, or partner's vasectomy) while on crenolanib and for 3 months following the last dose of crenolanib. Hormonal contraception alone is not an acceptable method of birth control for the purpose of this trial.
10. Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy and must agree to avoid to father a child (while on therapy and for 3 month after the last dose of crenolanib).
11. Willing to adhere to protocol specific requirements 12. Following receipt of verbal and written information about the study, the subject must provide signed informed consent before any study related activity is carried out. 13. Clinically significant toxic effects of prior therapy (expect hydroxyuria) resolved to Grade ≤ 1 before the start of study.

Exclusion Criteria

1. < 5% blasts in blood or marrow at screening, except if measurable extramedullary AML is confirmed
2. Acute promyelocytic leukemia (APL)
3. Known clinically active CNS leukemia
4. Clinically active or unstable graft-versus-host disease (GvHD) requiring treatment which precludes administration of chemotherapy as defined in this protocol
5. Prior anti-leukemia therapy within 14 days of enrollment for classical cytotoxic agents, and within 5x the half-life for other investigational agents

   * Prior use of hydroxyurea or isolated doses of cytarabine for palliation (i.e., control of WBC) are allowed but should be discontinued at least 24 hrs prior to enrollment.
   * Other agents used strictly with palliative intent might be allowed during this period after discussing with principal investigator
6. Pre-existing liver disease (e.g. cirrhosis, chronic hepatitis B or C, nonalcoholic steatohepatitis, sclerosing cholangitis)
7. Known HIV infection.
8. Evidence of ongoing, uncontrolled systemic infection or an uncontrolled local infection requiring therapy at the start of study.
9. "Currently active" second malignancy (other than non-melanoma skin cancer, carcinoma in situ of the cervix or prostatic intraepithelial neoplasia within 1 year). Subjects are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within 1 year.
10. Concurrent participation in another therapeutic clinical trial.
11. Pregnant or breastfeeding women
12. Subjects of childbearing potential not willing to use adequate contraception during study and 3 months after last dose of crenolanib
13. Subject with uncontrolled cardiac disease including congestive heart failure class III or IV by the NYHA, unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
14. Subject with concurrent severe and/or uncontrolled medical or psychiatric conditions that in the opinion of the investigator may impair the participation in the study or the evaluation of safety and/or efficacy
15. Inability to give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Arkansas, Little Rock, Arkansas
  - City of Hope Medical Center, Duarte, California
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: HAM Chemotherapy: Participants who had relapsed/refractory AML with FLT3 activating mutations who progressed on one prior chemotherapy received 100 mg crenolanib besylate tablets administered orally three times a day following HAM salvage chemotherapy.
- Arm B: FLAG-Ida Chemotherapy: Participants who had relapsed/refractory AML with FLT3 activating mutations who progressed on one prior chemotherapy received 100 mg crenolanib besylate tablets administered orally three times a day following FLAG-Ida salvage chemotherapy.
- Arm C: MEC Chemotherapy: Participants who had relapsed/refractory AML with FLT3 activating mutations who progressed on one prior chemotherapy received 100 mg crenolanib besylate tablets administered orally three times a day following MEC salvage chemotherapy.
Period: Overall Study
Arm/Group | Arm A: HAM Chemotherapy | Arm B: FLAG-Ida Chemotherapy | Arm C: MEC Chemotherapy
Started | 9 | 6 | 1
Completed | 6 | 4 | 1
Not Completed | 3 | 2 | 0
Not completed — Lack of Efficacy | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: HAM Chemotherapy | Arm B: FLAG-Ida Chemotherapy | Arm C: MEC Chemotherapy | Total
Number analyzed (Participants) | 9 | 6 | 1 | 16
Age, Continuous [Median (Full Range); unit: years] | 65 [36 to 78] | 66 [46 to 69] | 31 [31 to 31] | 65 [31 to 78]
Age, Customized [Count of Participants; unit: Participants]
  18 to 60 years | 2 | 2 | 1 | 5
  ≥ 60 years | 7 | 4 | 0 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 0 | 5
  Male | 5 | 5 | 1 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  White | 7 | 6 | 1 | 14
  Other | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 8 | 4 | 0 | 12
  Unknown | 0 | 0 | 0 | 0
ECOG [Count of Participants; unit: Participants] — ECOG performance status is graded by the investigator during a physical assessment. A greater ECOG grade is associated with greater impact of the disease on the ability of the subject to live. Grade 0 indicates subjects who are fully active and able to carry on all pre-disease performance. Grade 1 indicates subjects restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. Grade 2 indicates subjects who are ambulatory and capable of all selfcare but unable to carry out any work activities.
  Participants
    0 | 2 | 0 | 1 | 3
    1 | 5 | 5 | 0 | 10
    2 | 2 | 1 | 0 | 3
Antecedent Hematological Disorder [Count of Participants; unit: Participants] | 2 | 4 | 0 | 6
FLT3 Mutations [Count of Participants; unit: Participants] — Mutations in the gene encoding the trans-membrane tyrosine kinase FLT3. The type of FLT3 mutation detected by bone marrow assessment at diagnosis was collected. Subjects had either internal tandem duplications (ITD) in the juxtamembrane domain, point mutations or deletions in the tyrosine kinase domain (TKD) or both ITD and TKD mutations together.
  Participants
    ITD only | 3 | 0 | 1 | 4
    TKD only | 0 | 0 | 0 | 0
    ITD and TKD | 1 | 0 | 0 | 1
    FLT3 wildtype | 5 | 6 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to Crenolanib With Standard Salvage Chemotherapy
Description: To determine the response rate to crenolanib. Complete remission (CR) response criteria include a post-baseline bone marrow (BM) biopsy or aspiration % blasts <5%, absolute neutrophil count (ANC) >1×10^9/L and platelet count >100×10^9/L. CRi response included all CR criteria met, except participant did not have either platelet recovery or ANC recovery. CRh response included all CR criteria met, except subject only has partial platelet recovery and ANC recovery. Complete CR (CRc) response includes all subjects who achieve a CR, CRi and CRh. Partial Response (PR) response included a decrease of ≥50% in % blasts in the BM aspirate or biopsy from baseline but >5%. Morphologic Leukemia-Free State (MLFS) response included ≤5% in % blasts in the BM aspirate or biopsy.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: Participants who had relapsed/refractory AML with FLT3 activating mutations who progressed on one prior chemotherapy received 100 mg crenolanib besylate tablets administered orally three times a day following either HAM, MEC or FLAG-Ida salvage chemotherapy
Arm/Group | All Subjects | Arm A: HAM Chemotherapy | Arm B: FLAG-Ida Chemotherapy | Arm C: MEC Chemotherapy
Number analyzed (Participants) | 16 | 9 | 6 | 1
Participants
  Composite complete remission (CR+CRh+CRi) | 7 | 3 | 4 | 0
  MLFS | 3 | 2 | 0 | 1
  Clinical benefit (CRc+PR+MLFS) | 7 | 3 | 4 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30-days after the last dose, 1 year.
Groups:
- All Patients: Participants who had relapsed/refractory AML with FLT3 activating mutations who progressed on one prior chemotherapy received 100 mg crenolanib besylate tablets administered orally three times a day following standard salvage chemotherapy.
Arm/Group | All Patients | Arm A: HAM Chemotherapy | Arm B: FLAG-Ida Chemotherapy | Arm C: MEC Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/9 | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 6/16 | 4/9 | 2/6 | 0/1
Other Adverse Events (participants affected / at risk) | 16/16 | 9/9 | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=16) | Arm A: HAM Chemotherapy (N=9) | Arm B: FLAG-Ida Chemotherapy (N=6) | Arm C: MEC Chemotherapy (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 — Febrile neutropenia, Bacteraemia
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Upper gastrointestinal hemorrhage (General disorders) | 2 | 2 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Mental status change (Psychiatric disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=16) | Arm A: HAM Chemotherapy (N=9) | Arm B: FLAG-Ida Chemotherapy (N=6) | Arm C: MEC Chemotherapy (N=1)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 6 (6) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (10) | 5 (5) | 4 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 6 (6) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (7) | 4 (4) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Anal skin tags (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 2 (2) | 4 (4) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 2 (2) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 3 (3) | 2 (2) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 0 (0) | 4 (4) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood chloride increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT02626338/Prot_SAP_000.pdf